CLINICAL TRIAL: NCT03028909
Title: A Phase 2b, Randomized, Double-blind, Single-dose, Active-controlled, Dose Ranging Study to Evaluate the Efficacy and Safety of MEDI8852 in Adults Who Are Hospitalized With Influenza Caused by Type A Strains
Brief Title: Dose Ranging Study to Evaluate the Efficacy and Safety of MEDI8852 in Adults Who Are Hospitalized With Type A Influenza.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is withdrawn due to company decision.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6000C00003
Record Dates: First submitted 2016-12-06; First posted 2017-01-23 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2017-04

CONDITIONS: Influenza - Type A Strains
Keywords: Influenza A; MEDI8852
MeSH Terms: interventions — Oseltamivir; MEDI8852

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oseltamivir + low dose MEDI8852 (Experimental): Low Dose of MEDI8852 + Oseltamivir will be studied
  Interventions: Drug: Oseltamivir; Drug: MEDI8852
- Oseltamivir + high dose MEDI8852 (Experimental): High dose of MEDI8852 + Oseltamivir will be studied.
  Interventions: Drug: Oseltamivir; Drug: MEDI8852
- Oseltamivir + Placebo (Active Comparator): Oseltamivir in conjunction with placebo will be studied.
  Interventions: Drug: Oseltamivir; Drug: Placebo

INTERVENTIONS:
Drug: Oseltamivir — Standard of care for influenza caused by Type A strains
  Other Names: Tamiflu
Drug: MEDI8852 — MEDI8852 is a human IgG1 kappa monoclonal antibody (mAb) administered via infusion.
  Arms: Oseltamivir + high dose MEDI8852; Oseltamivir + low dose MEDI8852
Drug: Placebo — Salt-water solution containing no active ingredients.
  Arms: Oseltamivir + Placebo

SUMMARY:
The purposes of this study are to determine if MEDI8852 administered with standard of care (oseltamivir) will reduce the time to normalization of respiratory function for adults who are hospitalized with influenza caused by Type A strains and to determine if MEDI8852 has an acceptable safety profile in adults who are hospitalized with influenza caused by Type A strains.

DETAILED DESCRIPTION:
The MEDI8852 phase 2b study will evaluate the efficacy and safety of a single intravenous (IV) dose of MEDI8852 or placebo administered in conjunction with oseltamivir in adult subjects who are hospitalized with influenza caused by Type A strains. Approximately 450 subjects will be enrolled at study centers in North America, Europe, and other regions.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older at the time of screening. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act [HIPAA] in the United States, Data Privacy Directive in Europe) obtained from the subject/legal representative prior to performing any protocol related procedures, including screening evaluations.

Females of childbearing potential who are sexually active with a nonsterilized male partner must have evidence of not being pregnant upon enrollment and have a negative pregnancy test prior to administration of investigational product. Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), premenarchal, or postmenopausal (defined as 12 months with no menses without an alternative medical cause). Hospitalized ≤ 72 hours prior to receipt of a positive diagnostic test for influenza A; confirmed with positive rapid antigen test (supplied or approved by the sponsor), or confirmed with culture, polymerase chain reaction, or antigen testing at the study site. Onset of influenza symptoms ≤ 144 hours (≤ 6 days) prior to randomization. Receiving supplemental oxygen. Expected to participate in the study through Day 60.

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, would interfere with evaluation of study drugs or interpretation of subject safety or study results.
* Concurrent enrollment in another clinical study involving an investigational treatment. -Hospitalized > 72 hours (> 3 days) prior to receipt of a positive diagnostic test for influenza A.
* Receipt of > 72 hours or > 6 doses of treatment with a neuraminidase (NA) inhibitor. -Receipt of any investigational antiviral medications within 30 days prior to study drug dosing.
* Previous receipt of an influenza mAb within past 100 days.
* Pregnant or nursing female.
* History of allergic disease or reactions likely to be exacerbated by any components of the study drugs (MEDI8852 or oseltamivir).
* Diagnosis of influenza B infection within 14 days prior to randomization.
* Employees of the sponsor, clinical study site, or any other individuals involved with the conduct of the study, or immediate family members of such individuals.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-24 (Estimated); Primary Completion 2019-07-26 (Estimated); Study Completion 2019-07-26 (Estimated)

PRIMARY OUTCOMES:
Evaluation of efficacy as defined as time to normalization of respiratory function. | Through Day 14
  To evaluate the effect of MEDI8852 administered in conjunction with oseltamivir and the effect of oseltamivir alone in reducing time to normalization of respiratory function.
The occurence of Adverse Events | Through Day 28
  Occurrence of adverse events.
The occurence of Serious Adverse Events | Through Study Day 60
  Occurrence of serious adverse events.
The occurence of Adverse Events of Special Interest (AESIs) | Through Day 60
  Occurrence of Adverse Events of Special Interest.

SECONDARY OUTCOMES:
Assessment of the effect of MEDI8852 in reducing severity of clinical status. | Through Day 7
  Evaluation of the effect of MEDI8852 in reducing severity of clinical status defined by death, ICU, non-ICU hospitalization, but requiring supplemental oxygen, non-ICU hospitalization and not requiring supplemental oxygen, not hospitalized, but unable to resume normal activities, fully resumed normal activities
Evaluation of time to hospital discharge. | Through Day 60
  Evaluation of time to hospital discharge.
Quantitation of influenza viral shedding by qRT-PCR. | Through Day 60
  Evaluation of the effect of MEDI8852 in reducing the duration and quantity of viral shedding measured by qRT-PCR over time.
Evaluation of serum concentrations and PK of MEDI8852. | Through Day 60
  To evaluate serum concentration of MEDI8852 through Day 60.
Evaluation of serum ADA responses in serum through Day 60. | Through Day 60
  To evaluate the ADA response through Day 60.
Evaluation of time to ICU discharge. | Through Day 60
  Evaluation of time to ICU discharge.
Evaluation of the effect of MEDI8852 in reducing time to clinical resolution of individual vital sign abnormalities. | Through Day 14
  To evaluate time to clinical resolution of vital sign abnormalities.
Evaluation of Change in NEWS from baseline through Day 14. | Through Day 14
  To evaluate the effect of MEDI8852 in reducing NEWS.
Evaluation of the effect of MEDI8852 in reducing the duration of mechanical ventilation. | Through Day 60
  To evaluate duration of mechanical ventilation.
Evaluation of the effect of MEDI8852 in reducing the rates of ICU admission from the general ward. | Through Day 60
  To evaluate the rate of ICU admission from the general ward.
Evaluation to determine the effect of MEDI8852 on all-cause mortality | Through Day 60
  To evaluate All-cause mortality.
Evaluation of the effect of MEDI8852 on all-cause re-admission rates during the study. | Through Day 60
  To evaluate the rate of all-cause re-admission during the study.